CLINICAL TRIAL: NCT05637671
Title: Efficacy and Safety of Oxybutynin Versus Paroxetine in Breast Cancer Patients With Aromatase Inhibitor-induced Vasomotor Symptoms.
Brief Title: Efficacy and Safety of Oxybutynin Versus Paroxetine in Aromatase Inhibitor-induced Vasomotor Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa El-Sayed Mohammed Ahmed El-Sewiey, Teaching assistant, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL(3204)
Record Dates: First submitted 2022-11-12; First posted 2022-12-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Vasomotor Symptoms
Keywords: Hot flashes; vasomotor symptoms; oxybutynin; paroxetine; aromatase inhibitors; breast cancer
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oxybutynin (Active Comparator): One study group will receive 10 mg of oxybutynin ER orally once daily for 12 weeks
  Interventions: Drug: oxybutynin ER
- paroxetine (Active Comparator): the other group will receive 12.5 mg of paroxetine CR orally once daily for 12 weeks
  Interventions: Drug: Paroxetine CR

INTERVENTIONS:
Drug: oxybutynin ER — One study group will receive 10 mg of oxybutynin ER orally once daily for 12 weeks.
  Arms: oxybutynin
Drug: Paroxetine CR — the other group will receive 12.5 mg of paroxetine CR orally once daily for 12 weeks.
  Arms: paroxetine

SUMMARY:
Breast cancer is the most prevalent cancer type worldwide. In Egypt, It is the second most common type of cancer and the most common one in women with about 22 thousand new cases in 2020. Around 70% of newly diagnosed patients are hormone receptor-positive and, unfortunately, the disease is often diagnosed at the advanced stage.

In postmenopausal women with hormone receptor-positive breast cancer, aromatase inhibitors (AIs) are the first-line adjuvant therapy according to National Comprehensive Cancer Network (NCCN) guidelines. Although, they showed superiority in efficacy to tamoxifen in this type of breast cancer, one of the most annoying adverse effects of the aromatase inhibitors are the vasomotor symptoms. They could be as severe as the patient would prefer discontinuing the medication. The underlying mechanism responsible for those adverse effects is that AIs suppress plasma estrogen levels by inhibiting the enzyme responsible for the conversion of androgens to estrogens in peripheral tissues. This estrogen depletion has been linked to an increase in hot flushes by decreasing endorphin levels and increasing that of norepinephrine and serotonin, followed by instability of the hypothalamic thermoregulatory set point which allows changes in the body temperature and in hot flash sensation.

Hormone replacement therapy is considered first-line treatment for vasomotor symptoms. However, it is not preferred to be used in breast cancer patients especially those with hormone receptor positive breast cancer. So, many drugs have been investigated for their efficacy in reducing the frequency and severity of vasomotor symptoms. The only FDA-approved drug to treat moderate-to-severe vasomotor symptoms is paroxetine. Paroxetine is a selective serotonin reuptake inhibitor (SSRI) which is used mainly in major depressive disorder and other psychiatric conditions like anxiety disorders. It has proved an efficacy in reducing frequency and severity of hot flushes in post-menopausal women. But, there are several concerns regarding its use with tamoxifen in breast cancer patients. There is a competition between paroxetine and tamoxifen for hepatic CYP2D6, so, paroxetine prevents conversion of tamoxifen into its active metabolite.

Oxybutynin has shown efficacy in relieving vasomotor symptoms. Oxybutynin is an anticholinergic used usually in urinary incontinence. It has an advantage over other SSRIs that it lacks the interaction with tamoxifen on CYP2D6 and, therefore, with the anticancer effect of tamoxifen treatment in breast cancer patients.

To our knowledge, there are no head-to-head studies comparing the efficacy and safety of paroxetine versus oxybutynin in reducing frequency and severity of vasomotor symptoms especially in breast cancer patients taking aromatase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal female patients who are 18 years of age or older.
2. Patients diagnosed with hormone receptor-positive breast cancer stage 0 - IIIC (non-advanced breast cancer) who are taking aromatase inhibitors as adjuvant therapy (post-surgery) and having Significant vasomotor symptoms, defined as a mean of 5 moderate to severe hot flashes per day.
3. Have an Eastern Cooperative Oncology Group performance status rating (ECOG-PSR) ˂ 2.
4. Life expectancy greater than 6 months.
5. Normal serum creatinine level and bilirubin level is less than two times the normal level.
6. Serum follicle-stimulating hormone (FSH) levels above 40 mIU/mL.

Exclusion Criteria:

1. Patients taking tamoxifen as adjuvant therapy.
2. Metastatic breast cancer.
3. Other treatments used for hot flashes, antidepressants, and monoamine oxidase inhibitors (except if they are discontinued for at least one month before study entry).
4. Hypersensitivity to paroxetine or oxybutynin.
5. Presence of a condition requiring use of an anticholinergic agent.
6. Untreated hypertension.
7. Impaired liver or kidney function.
8. Unstable cardiac disease.
9. Pregnancy or breastfeeding.
10. History of self-injurious behavior.
11. History of clinical diagnosis or treatment of any psychiatric disorder.
12. Prior use of oxybutynin or paroxetine for hot flushes.
13. Recent use of oxybutynin or paroxetine for conditions other than vasomotor symptoms unless they are stopped at least 30 days before the study entry.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 146 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of oxybutynin compared to paroxetine through hot flashes diary | 12 weeks
  Comparing the efficacy of oxybutynin to paroxetine in reducing frequency and severity of moderate to severe vasomotor symptoms in breast cancer patients receiving aromatase inhibitors using hot flashes diary.
Efficacy of oxybutynin compared to paroxetine through The Pittsburgh Sleep Quality Index questionnaire | 12 weeks
  Comparing the efficacy of oxybutynin to paroxetine in reducing sleep disturbances in breast cancer patients receiving aromatase inhibitors using The Pittsburgh Sleep Quality Index questionnaire.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 weeks
  Comparing the safety of oxybutynin to paroxetine through an every-other-week assessment of possible adverse events (dry mouth, dyspepsia, diarrhea, constipation, urinary tract infections, suicidal ideation, fatigue, headache, dizziness, etc.).
Safety of oxybutynin compared to paroxetine on kidney through serum creatinine assessment | 12 weeks
  Comparing the safety of oxybutynin to paroxetine on kidney through assessment of serum creatinine abnormalities on week 12 compared to baseline.
Safety of oxybutynin compared to paroxetine on kidney through blood urea nitrogen assessment | 12 weeks
  Comparing the safety of oxybutynin to paroxetine on kidney through assessment of blood urea nitrogen abnormalities on week 12 compared to baseline.
Safety of oxybutynin compared to paroxetine on liver through Alanine aminotransferase assessment | 12 weeks
  Comparing the safety of oxybutynin to paroxetine through assessment of Alanine aminotransferase abnormalities on week 12 compared to baseline.
Safety of oxybutynin compared to paroxetine on liver through aspartate aminotransferase assessment | 12 weeks
  Comparing the safety of oxybutynin to paroxetine through assessment of aspartate aminotransferase abnormalities on week 12 compared to baseline.
Safety of oxybutynin compared to paroxetine on liver through bilirubin assessment | 12 weeks
  Comparing the safety of oxybutynin to paroxetine through assessment of bilirubin abnormalities on week 12 compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Dar El-Salam Cancer Hospital, Cairo, Governorate, Egypt